CLINICAL TRIAL: NCT00296660
Title: Acute HIV-1 Infection Prospective Cohort Study
Brief Title: Acute HIV Infection Observational Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CHAVI 001
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: Acute Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- 1: Proven acute HIV-1 infection
- 1A: Sexual partners of members of Group 1
- 2: Established HIV-infection
- 3: HIV-1 uninfected

SUMMARY:
The purpose of this study is to collect data and body fluid samples from people with acute or established HIV infection and from HIV uninfected people. Data from this study will be used to better understand properties of HIV, including HIV transmission and the differences between acute and established HIV infections.

DETAILED DESCRIPTION:
Previous studies have identified strategies for the large-scale identification of acute HIV infections. One system using such strategies has already been implemented in North Carolina, and this system will be used in this study run by the Center of HIV/AIDS Vaccine Immunology (CHAVI). This study will collect data on the mechanism of HIV transmission and the genetic, biologic, antigenic, and structural characteristics of the virus. The study will enroll HIV infected people with acute HIV infection and their sexual partners, people with established HIV infection, and HIV uninfected people.

This study will last 96 weeks. Group 1 participants will be people with acute HIV infection. These participants will have 15 study visits; some visits will include a physical exam and medical history. Group 1 will also be asked to complete a sexual behavioral assessment at study entry and every 12 weeks thereafter. Group 2 participants will be people with established HIV infection. Group 3 participants will be HIV uninfected people. Groups 2 and 3 will have 10 study visits; some visits will include a physical exam and medical history. Groups 2 and 3 will also be asked to complete a sexual behavioral assessment at study entry, every 12 weeks until Week 72, and Week 96. Group 3 will undergo HIV testing at each visit and will receive pre- and post-test counseling.

At each visit, participants will undergo HIV safe sex counseling and will update their locator information. Blood, genital secretion, and breast milk collection will also occur at each visit.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Willing to receive HIV test results
* Willing to provide updated locator information during the study

Inclusion Criteria for Group 1:

* Acute HIV infection OR sexual partner of a Group 1 participant with acute HIV infection

Inclusion Criteria for Group 2:

* Established HIV infection (positive HIV antibody test and positive HIV Western blot)

Inclusion Criteria for Group 3:

* HIV uninfected

Exclusion Criteria for All Participants:

* Plan to relocate out of the area during the study or have a job or other obligations that may require long absences from the area
* Currently on antiretroviral therapy. Women who previously took antiretroviral therapy for the prevention of mother-to-child transmission of HIV are not excluded.
* Any other condition that, in the opinion of the investigator, may interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 1300 with either an acute HIV-1 infection, established HIV-1 infection, or without HIV-1 infection will be enrolled. Sexual partners of those with an acute infection will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2006-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of acute HIV infection | Throughout study
Characteristics of transmitted virus in acute HIV infection | Throughout study
Immune responses contributing to viral control and/or protection against HIV infection | Throughout study
Genetic factors contributing to early virus control and/or protection from HIV infection | Throughout study
Clinical, laboratory, and behavioral characteristics of individuals at diverse sites with acute HIV infection and their sexual partners, and appropriate controls | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Myron S. Cohen, MD, Study Chair — Medicine, Microbiology, and Immunology and Public Health, Division of Infectious Diseases, University of North Carolina Center for Infectious Diseases
Locations (9):
- United States (2):
  - UNC School of Medicine, Div. of Infectious Diseases CHAVI CRS, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr., Infectious Diseases Clinic CHAVI CRS, Durham, North Carolina
- Malawi (2):
  - Queen Elizabeth Hosp., Malawi College of Medicine-Johns Hopkins Research Project CHAVI CRS, Blantyre
  - Kamuzu Central Hosp. CHAVI CRS, Lilongwe
- South Africa (3):
  - Univ. of Witwatersrand, Chris Hani Baragwanath Hosp., Reproductive Health Research Unit CHAVI CRS, Johannesburg, Gauteng
  - CAPRISA eThekwini CHAVI CRS, Durban, KwaZulu-Natal
  - Aurum Institute for Health Research CHAVI CRS, Klerksdorp
- Kilimanjaro Christian Med. Ctr. CHAVI CRS, Moshi, Tanzania
- Uganda Virus Research Institute, MRC/UVRI Uganda Research Unit on AIDS CHAVI CRS, Entebbe, Uganda

REFERENCES:
- [Background] Lindback S, Thorstensson R, Karlsson AC, von Sydow M, Flamholc L, Blaxhult A, Sonnerborg A, Biberfeld G, Gaines H. Diagnosis of primary HIV-1 infection and duration of follow-up after HIV exposure. Karolinska Institute Primary HIV Infection Study Group. AIDS. 2000 Oct 20;14(15):2333-9. doi: 10.1097/00002030-200010200-00014. PMID 11089621
- [Background] Pilcher CD, Eron JJ Jr, Galvin S, Gay C, Cohen MS. Acute HIV revisited: new opportunities for treatment and prevention. J Clin Invest. 2004 Apr;113(7):937-45. doi: 10.1172/JCI21540. PMID 15057296
- [Background] Pilcher CD, Fiscus SA, Nguyen TQ, Foust E, Wolf L, Williams D, Ashby R, O'Dowd JO, McPherson JT, Stalzer B, Hightow L, Miller WC, Eron JJ Jr, Cohen MS, Leone PA. Detection of acute infections during HIV testing in North Carolina. N Engl J Med. 2005 May 5;352(18):1873-83. doi: 10.1056/NEJMoa042291. PMID 15872202
- [Background] Pilcher CD, McPherson JT, Leone PA, Smurzynski M, Owen-O'Dowd J, Peace-Brewer AL, Harris J, Hicks CB, Eron JJ Jr, Fiscus SA. Real-time, universal screening for acute HIV infection in a routine HIV counseling and testing population. JAMA. 2002 Jul 10;288(2):216-21. doi: 10.1001/jama.288.2.216. PMID 12095386
- [Background] Soogoor M, Daar ES. Primary human immunodeficiency virus type 1 infection. Curr HIV/AIDS Rep. 2005 Jun;2(2):55-60. doi: 10.1007/s11904-005-0019-1. PMID 16091249